CLINICAL TRIAL: NCT01665976
Title: A Single Center, Randomized, Single Dose, Open-label, Four Period Cross-over Study to Investigate the Relative Bioavailability of RO4917838 and the Effect of Food Following Oral Administration in Healthy Subjects
Brief Title: A Study of the Relative Bioavailability of Single Dose RO4917838 and the Effect of Food in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BP25593; 2012-000739-13 (EudraCT Number)
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (4):
- A: film coated tablets, fasted condition (Experimental)
  Interventions: Drug: RO4917838
- B: film coated tablets, fed condition (Experimental)
  Interventions: Drug: RO4917838
- C: hard gelatin capsules (Experimental)
  Interventions: Drug: RO4927838
- D: oral suspension (Experimental)
  Interventions: Drug: RO4917838

INTERVENTIONS:
Drug: RO4917838 — film coated tablet, single dose
  Arms: A: film coated tablets, fasted condition; B: film coated tablets, fed condition
Drug: RO4917838 — oral suspension, single dose
  Arms: D: oral suspension
Drug: RO4927838 — hard gelatin capsule, single dose
  Arms: C: hard gelatin capsules

SUMMARY:
This single center, randomized, single dose, open-label, four period cross-over study will evaluate the relative bioavailability of RO4917838 and the effect of food following oral administration in healthy volunteers. Subjects will receive in randomized order single oral doses of RO4917838 film coated tablets, either in the fasted or fed condition, or RO4917838 hard gelatin capsules or RO4917838 oral suspension, with a washout period of at least 21 days between treatments. Anticipated time on study will be up to 23 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, 18 to 65 years of age, inclusive
* Body mass index (BMI) 18 to 30 kg/m2 inclusive
* Healthy as determined by the Investigator on the basis of medical and surgical history and a complete physical examination
* Non-smoker or smoker of fewer than 10 cigarettes per day; subject must be able to refrain from smoking during the in-patient stays
* Females who are not postmenopausal or surgically sterile must agree to use two adequate methods of contraception as defined by protocol during the treatment period and for at least one month after the last dose of study drug

Exclusion Criteria:

* Any condition or disease detected during the medical interview/physical examination that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the Investigator
* History of alcoholism, drug abuse and/or drug addiction within the last year prior to Period 1. Day -1 of the study
* History of any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, allergic, dermatologic, hematologic, neurologic, psychiatric disease, or cancer
* Any history of depressive episodes or treatment with antidepressants
* Any significant allergic reactions against any drug, or multiple allergies in the judgement of the Investigator
* Pregnant or lactating females
* Positive for hepatitis B, hepatitis C or HIV infection
* Participation in another investigational study of any type within 90 days of RO4917838 administration or within 6 times the elimination half-life of the tested drug, whichever is longer

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Effect of high fat and high caloric food on the relative bioavailability of single dose RO4917838 film coated tablets (FCT): Area under the concentration-time curve (AUC) | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 h post-dose, and up to Day 12
Relative bioavailability of single dose RO4917838 hard gelatin capsules as compared to FCT: Area under the concentration-time curve | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 h post-dose, and up to Day 12
Relative bioavailability of single dose RO4917838 oral suspension as compared to FCT | Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 h post-dose, and up to Day 12

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Rueil-Malmaison, France